CLINICAL TRIAL: NCT04570501
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled Study of the Safety and Efficacy of Angiotensin (1-7) for the Treatment of COVID-19 in Hospitalized Patients
Brief Title: Angiotensin (1-7) for the Treatment of COVID-19 in Hospitalized Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinuation of drug candidates
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58189
Record Dates: First submitted 2020-09-28; First posted 2020-09-30 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Angiotensin (1-7) (Experimental): Participants receive treatment for 7 days.
  Interventions: Drug: Angiotensin-(1-7)
- Placebo (Placebo Comparator): Participants receive treatment for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Angiotensin-(1-7) — Ang (1-7) administered by continuous intravenous (IV) infusion
  Arms: Angiotensin (1-7)
Drug: Placebo — Placebo (normal saline) administered by continuous intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the safety and efficacy of intravenous (IV) infusion of Ang (1-7) compared to placebo with respect to time to recovery, disease severity, need for mechanical ventilation or extracorporeal membrane oxygenation (ECMO), and mortality in patients with COVID 19.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms suggestive of COVID-19 infection including cough or dyspnea
* Laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) test ≤7 days before randomization
* Currently hospitalized or in an emergency department with planned hospitalization
* Peripheral capillary oxygen saturation (SpO2) ≤93% on room air or partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) <300 at Screening

Exclusion Criteria:

* Simultaneous participation in any other clinical study incompatible with this one
* Treatment with an antibody immunotherapy that is not standard of care for COVID-19 within 4 weeks of Screening
* Requirement for mechanical ventilation or ECMO at Screening
* Hypotension at Screening, defined as supine BP <95 mm Hg systolic or <55 mm Hg diastolic
* Severe liver injury defined as AST or ALT ≥5x the upper limit of normal
* Severe kidney failure defined as an estimated glomerular filtration rate (eGFR) <30 mL/min
* Any known immune deficiency
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | Up to 29 days
  Time to recovery, defined as attaining a score of 6, 7, or 8 on the COVID-19 disease severity scale, an 8 point ordinal scale used in the NIH Adaptive COVID-19 Treatment Trial (ACTT; NCT04280705).
  1. = Death;
  2. = Hospitalized and on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  3. = Hospitalized and on non-invasive ventilation or high-flow oxygen devices;
  4. = Hospitalized and requiring supplemental oxygen;
  5. = Hospitalized and not requiring supplemental oxygen but requiring ongoing medical care (COVID-19-related or otherwise);
  6. = Hospitalized and not requiring supplemental oxygen and no longer requiring ongoing medical care;
  7. = Not hospitalized, limitation on activities and/or requiring home oxygen;
  8. = Not hospitalized, no limitation on activities

SECONDARY OUTCOMES:
Incidence of mortality at Day 29 | 29 days
Number of days alive and not on mechanical ventilator or ECMO in the 28 days following first dose | Up to 29 days
Number of participants requiring mechanical ventilation or ECMO, or dying, through Day 29 | Up to 29 days
COVID-19 disease severity scale score on Day 8 | Day 8
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
COVID-19 disease severity scale score on Day 15 | Day 15
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
COVID-19 disease severity scale score on Day 22 | Day 22
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).
COVID-19 disease severity scale score on Day 29 | Day 29
  COVID-19 disease severity scale (range; 1-8, higher scores correspond to better health state).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin V Grimes, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No